CLINICAL TRIAL: NCT04928300
Title: Diaphragmatic Function, Pain Quality & Anti-inflammatory Properties: A Low Dose Dexmedetomidine Versus Ketamine in Patients With Multiple Fracture Ribs Needing Conservative Treatment
Brief Title: Low Dose Dexmedetomidine Versus Normal Saline in Multiple Fracture Ribs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300614
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): Dexmedetomidine infusion IV for 5 days.
  Interventions: Drug: Dexmedetomidine
- Group C (Placebo Comparator): The same dose and duration of normal saline will be given.
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — low dose dexmedetomidine infusion 0.2 µ/kg/hour IV for 5 days.
  Other Names: Precedex
  Arms: Group D
Other: 0.9% saline — the same dose and duration of normal saline will be given for 5 days.
  Other Names: Normal saline
  Arms: Group C

SUMMARY:
In our study, we assess the diaphragmatic function, pain quality and anti-inflammatory properties between low dose infusion of dexmedetomidine normal saline in patients with multiple fracture ribs on conservative treatment.

DETAILED DESCRIPTION:
A written informed consent from patients or thier legal guardians, Patients will be assigned randomly to two groups (30 subjects each) with traumatic multiple fracture ribs 3 ribs or more. After thoracic epidural is inserted, the drug study intervention will be started and run for 5 days during ICU admission. In (Group D) low dose dexmedetomidine infusion 0.2 µ/kg/hour IV for 5 days. In (Group C) the same dose and duration of normal saline will be given.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-65 years) of American Society of Anaesthesiologists (ASA) physical status I-II
* Traumatic multiple fracture ribs 3 ribs or more, who will be subjected to thorough assessments including chest 3D-CT
* Undergoing conservative treatment (chest strappings)
* Intractable pain with visual analogue scale (VAS) over 6 after traditional therapies
* Glasgow Coma Scale (GCS) ≥ 13.

Exclusion Criteria:

* Multiple traumas to body parts other than chest with an abbreviated injury scale over 3
* Serious head trauma with a Glasgow coma scale lower than 13
* Mechanically ventilated patients
* Massive hemothorax
* Injury to the trachea or bronchus with requirement for immediate surgery
* Dementia
* Use of corticosteroids during ICU stay
* Sepsis
* Continued use of neuromuscular blocking agents and aminoglycosides antibiotic use as they are known risk factors for ICU-acquired weakness and any known hypersensitivity
* Contraindication to the study drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic diaphragm function | 5 days
  Diaphragmatic excursion and thickness will be assessed by ultasound for 5 days with diaphragmatic dysfunction (DD) is diagnosed if diaphragmatic excursion is <10 mm and diaphragmatic thickness is <2 mm. .

SECONDARY OUTCOMES:
Visual analogue scale for pain | 48 hours
  Severity of pain will be assessed and scored by 10-point visual analogue scale (VAS). The patients will be instructed on how to use VAS for the assessment of the degree of pain (with 0 representing no pain and 10 cm representing the worst imaginable pain). According to the degree pain given by the patient, classification of pain severity will be done as follows: no pain = 0, mild pain <3, moderate pain 4-6 and severe pain >7. VAS will be recorded at zero time before drug intervention, 4 h, 6 h, 12 h, 24 h and 48 h after the start of the treatment in all groups by the anesthesia resident not involved in any other part of the study.

OTHER OUTCOMES:
Neutrophil/lymphocyte ratio (NLR) | 3 days
  From complete blood picture, neutrophil/lymphocyte ratio is measured to assess anti-inflammatory properties of the study drugs daily for 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bossolasco M, Bernardi E, Fenoglio LM. Continuous serratus plane block in a patient with multiple rib fractures. J Clin Anesth. 2017 May;38:85-86. doi: 10.1016/j.jclinane.2016.12.015. Epub 2017 Jan 30. No abstract available. PMID 28372691